CLINICAL TRIAL: NCT07150585
Title: The Influence of Irrigation Activation Systems on Postoperative Pain and Periapical Lesion Healing in Single-visit Root Canal Retreatment Cases: A Randomized Clinical Trial
Brief Title: Effects of Irrigation Activation Systems on Postoperative Pain and Lesion Healing in Single-Visit Retreatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Burcu Serefoglu, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUDF-ETK- 24-3/86; EU-GAP-32275 (Other Grant/Funding Number: Ege University)
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Retreatment; Asymptomatic Apical Periodontitis
Keywords: Er:YAG laser; Irrigation activation; Postoperative pain; Sonic irrigation; Ultrasonic irrigation; Single-visit; Nonsurgical endodontic retreatment; outcome of nonsurgical retreatment; periapical lesion healing
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasonic Activation Group (Active Comparator): In the group where passive ultrasonic activation was applied to enhance the efficacy of the final irrigation protocol, an Ultra X device (Eighteeth, Changzhou Sifary Medical Technology Co., Ltd.) equipped with silver 21 mm, 0.2-taper irrigation tips was used. The tip was positioned 2 mm short of the working length and moved in an up-and-down motion to activate 17% EDTA for three 20-second cycles (3 × 2 mL), followed by 2.5% NaOCl for three identical cycles
  Interventions: Device: Ultrasonic Activation Group
- Sonic Activation Group (Active Comparator): In the sonic activation group, a polyamide 20 mm, 0.05 taper EDDY tip (VDW, Munich, Germany) mounted on a sonic air scaler (TA 200, Micron, Japan) was used to enhance the efficacy of the final irrigation protocol. The tip was inserted 2 mm short of the working length and agitated in an up-and-down motion to activate 17% EDTA for three 20-second cycles (3 × 2 mL), followed by 2.5% NaOCl for three identical cycles.
  Interventions: Device: Sonic Activation Group
- Laser Activation Group (Active Comparator): In the laser group, an Er:YAG Lightwalker device (Fotona, Ljubljana, Slovenia) in Shock Wave Enhanced Emission Photoacoustic Streaming (SWEEPS) mode (2940 nm, 20 mJ, 15 Hz, 0.3 W, 25 μs pulse duration) was used. A SWEEPS fiber tip mounted on the H14 handpiece was positioned in the access cavity with air and water pressures set to zero, and was used to activate 17% EDTA for three 20-second cycles (3 × 2 mL), followed by 2.5% NaOCl for three identical cycles.
  Interventions: Device: Laser Activation Group

INTERVENTIONS:
Device: Ultrasonic Activation Group — In this group, during single-visit nonsurgical root canal retreatment, irrigant activation in the final irrigation protocol was performed using the Ultra X device (Eighteeth) with ultrasonic tips.
  Other Names: (Ultra X,Eighteeth)
  Arms: Ultrasonic Activation Group
Device: Sonic Activation Group — In this group, during single-visit nonsurgical root canal retreatment, irrigant activation in the final irrigation protocol was performed using an EDDY sonic activation tip (VDW, Munich, Germany)
  Other Names: (EDDY,VDW)
  Arms: Sonic Activation Group
Device: Laser Activation Group — In this group, during single-visit nonsurgical root canal retreatment, irrigant activation in the final irrigation protocol was performed using the LightWalker (Fotona, Ljubljana, Slovenia) Er:YAG laser device in SWEEPS mood
  Other Names: (Lightwalker AT,Fotona)
  Arms: Laser Activation Group

SUMMARY:
In this superiority randomized clinical trial with a parallel design, 75 asymptomatic maxillary anterior teeth with 2-5 mm periapical lesions and a history of primary root canal treatment (PRCT) at least four years earlier were included. Patients were randomly assigned, using a randomization sequence generated on www.random.org, and divided into three groups. In all patients, existing canal fillings were removed using Remover rotary file (Coltene, MicroMega) and hand files. Working lengths were determined with an apex locator and canals reshaped using the step-back technique. For the final irrigation, side-vented needles were positioned 2 mm short of the working length. Activation was performed with Ultra X (Eighteeth) in the ultrasonic group, EDDY (VDW) in the sonic group, and an Er:YAG laser (LightWalker, Fotona) in SWEEPS mode (2940 nm, 5 μs, 20 mJ, 15 Hz) in the laser group. In all groups, each irrigant (EDTA followed by NaOCl) was activated in three cycles of 20 seconds. All canals were obturated with gutta-percha and a bioceramic sealer, and restored with composite. Pain levels were recorded using the Visual Analog Scale (VAS) 0, 6, 12, 24, 48, and 72 hours, and on day 7. The completed forms were collected by another independent investigator blinded to the group assignments. At the end of the treatment, periapical radiographs were obtained and recorded from all patients. Patients whose treatment was completed will be recalled at the 6th, 12th, and 24th months for follow-up periapical radiographs, and the comparison of healing among the groups will be evaluated as a secondary outcome based on changes in the PAI index.

DETAILED DESCRIPTION:
This randomized controlled trial, employing a double-blind, single-center, parallel-group superiority design, was conducted and reported in line with the Preferred Reporting Items for Randomized Trials in Endodontics (PRIRATE) 2020 guidelines. Ethical approval was obtained from the Ege University Clinical Research Ethics Committee, Izmir, Turkey (Approval No: 24-3/86). Participant recruitment took place at the Department of Endodontics, Ege University Faculty of Dentistry, between December 2024 and June 2025. Prior to inclusion, all participants received verbal and written information about the study's objectives, procedures, potential benefits, and risks, and provided signed informed consent. Sample-size estimation was based on postoperative pain on the VAS as the primary outcome. Using G*Power 3.1.9.6 for a repeated-measures ANOVA (between-within interaction; three groups; seven time points), with α=0.05, power=95%, and an effect size f=0.358, the required total sample size was 75 (n=25 per group; allocation ratio 1:1:1). Medically healthy individuals aged 18-65 who agreed to participate and attend follow-up visits were enrolled in this randomized controlled trial. Only asymptomatic maxillary anterior teeth with completed root development, a history of root canal treatment performed at least four years earlier, and periapical lesions measuring 2-5 mm, with healthy periodontal status and no mobility, were included. Patients with systemic disease, pregnancy, or known allergies to treatment materials, as well as teeth presenting symptoms, lesions smaller than 2 mm or larger than 5 mm, open apices, advanced periodontal disease, or mobility, were excluded. All treatment procedures were performed by a single operator (B.G.), with two years of clinical practice in the endodontics department. Under rubber dam isolation, existing restorations and carious lesions, if present, were removed. Previous root canal fillings were removed using a rotary Remover file (Coltene MicroMega, Besançon, France) and a Hedström file (Dentsply Maillefer, Ballaigues, Switzerland). Due to the passive tip design of the Remover file, a retention space of 1-2 mm was first created within the filling material using a #3 Gates-Glidden drill. The Remover file was used with an X-Smart Plus endodontic motor (500 rpm, 2.5 Ncm) in 3 mm strokes to remove filling material from the coronal and middle thirds. The remaining 3 mm of filling material in the apical third was removed using a Hedström hand file of a size corresponding to the tooth's apical diameter. Working length was determined with an apex locator (RayPex 6, VDW, Munich, Germany) and canals reshaped using the step-back technique. Between each file change, canals were irrigated using a 30-gauge irrigation needle (Kerr Hawe Sa, Bioggio, Switzerland) with 2 mL of 2.5% sodium hypochlorite (NaOCl) (Wizard, Rehber Kimya, Turkey) and 2 mL of 17% ethylenediaminetetraacetic acid (EDTA) (Sigma Chemical Co., St. Louis, MO, USA). In total, 20 mL of NaOCl and 8-10 mL of EDTA were used during the removal and reshaping procedures for each tooth. The master gutta-percha cone of the determined apical size was fitted to the working length until tug-back was achieved, and a periapical radiograph was taken for confirmation. The sequence of the final irrigation protocol for each patient was pre-assigned at the start of the study using the automated randomization method available at www.random.org. Allocation was concealed until this stage to maintain blinding. In the ultrasonic group, an Ultra X device (Eighteeth, Changzhou Sifary Medical Technology Co., Ltd.) equipped with silver 21 mm, 0.2-taper irrigation tips was used. The tip was positioned 2 mm short of the working length and moved in an up-and-down motion to activate 17% EDTA for three 20-second cycles (3 × 2 mL), followed by 2.5% NaOCl for three identical cycles. In the sonic group, a polyamide EDDY tip (20 mm, 0.05 taper; VDW, Munich, Germany) was mounted on a sonic air scaler (TA 200, Micron, Japan). The tip was inserted 2 mm short of the working length and agitated in an up-and-down motion, activating 17% EDTA for three 20-second cycles (3 × 2 mL), followed by 2.5% NaOCl for three identical cycles. In the laser group, an Er:YAG Lightwalker device (Fotona, Ljubljana, Slovenia) in Shock Wave Enhanced Emission Photoacoustic Streaming (SWEEPS) mode (2940 nm, 20 mJ, 15 Hz, 0.3 W, 25 μs pulse duration) was used. A SWEEPS fiber tip mounted on the H14 handpiece was positioned in the access cavity with air and water pressures set to zero, and irrigation activation was performed in the same manner as in the other two groups. Canals were finally rinsed with 5 mL of distilled water and dried with paper points. Root canal obturation was then performed using the master cone gutta-percha (Diadent Group International Inc., South Korea) and BioRoot RCS sealer (Septodont, France) with the lateral compaction technique. The canal orifices were sealed with a 3-mm layer of flowable composite (RubyFlow, Rubydent) and the coronal restorations were completed with resin composite (Solare X, GC). Final radiographs were taken using a parallel film holder to ensure the same positioning as the initial periapical images. Patients whose treatment was completed will be recalled at the 6th, 12th, and 24th months for follow-up periapical radiographs, and the comparison of healing among the groups will be evaluated as a secondary outcome based on changes in the PAI index.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients
* Patients between 18 and 65 years of age
* Patients with previously root canal-treated teeth who are asymptomatic
* Patients with maxillary anterior teeth presenting with periapical lesions measuring between 2-5 mm
* Teeth with completed root development and healthy periodontal status
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients with any systemic disease
* Pregnant patients
* Patients with allergies to the materials used during the procedure
* Patients with previously root canal-treated teeth who are symptomatic
* Teeth in the maxillary anterior region with periapical lesions smaller than 2 mm or larger than 5.1 mm
* Teeth with open apices
* Teeth with advanced periodontal disease and mobility
* Patients who did not consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain | From immediately after retreatment to 7 days postoperatively
  Following single-visit nonsurgical root canal retreatment performed with different irrigation activation techniques, the Visual Analog Scale (VAS) was used to assess and compare the patients' pain levels, and the patients were instructed to record their pain at 0, 6, 12, 24, 48, and 72 hours, as well as on the 7th day. Patients were informed that a score of 0 represented no pain, while a score of 10 represented the maximum pain, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Radiographic healing of periapical lesions | At 6, 12, and 24 months after retreatment
  Following single-visit nonsurgical root canal retreatment performed with different irrigation activation techniques, the Periapical Index (PAI) was used to evaluate and compare periapical lesion healing. Patients will be recalled at 6, 12, and 24 months post-treatment for radiographic examinations. PAI scores range from 1 to 5, where 1 indicates a healthy periapical status and 5 represents severe periapical pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Department of Endodontics, Izmır, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mittal N, Baranwal HC, Gupta S, Shankari T, Gupta S, Kharat S. Comparative analysis of reduction in pain scores after single visit root canal treatment using endodontic irrigation protocols, namely, Conventional needle irrigation, PUI, PIPS and SWEEPS: A randomized control trial. J Conserv Dent. 2023 Mar-Apr;26(2):143-149. doi: 10.4103/jcd.jcd_450_22. Epub 2023 Mar 16. PMID 37205889
- [Background] Liapis D, De Bruyne MAA, De Moor RJG, Meire MA. Postoperative pain after ultrasonically and laser-activated irrigation during root canal treatment: a randomized clinical trial. Int Endod J. 2021 Jul;54(7):1037-1050. doi: 10.1111/iej.13500. Epub 2021 Mar 9. PMID 33595920
- [Background] Erkan E, Gundogar M, Uslu G, Ozyurek T. Postoperative pain after SWEEPS, PIPS, sonic and ultrasonic-assisted irrigation activation techniques: a randomized clinical trial. Odontology. 2022 Oct;110(4):786-794. doi: 10.1007/s10266-022-00700-0. Epub 2022 Mar 10. PMID 35267110